CLINICAL TRIAL: NCT00448630
Title: A MULTI-CENTER, NON-INVASIVE OBSERVATIONAL STUDY OF METABOLIC SYNDROME PARAMETERS IN SCHIZOPHRENIC PATIENTS USING ATYPICAL ANTIPSYCHOTICS
Brief Title: An Observational Study On Metabolic Syndrome Parameters In Schizophrenia Patients Treated With Atypical Antipsychotics
Acronym: MESSAGE
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1281160
Record Dates: First submitted 2007-03-16; First posted 2007-03-19 (Estimated); Results first posted 2010-07-07 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia; Metabolic Syndrome X
Keywords: Atypical antipsychotics; Metabolic syndrome; Safety
MeSH Terms: conditions — Schizophrenia; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood (fasting blood glucose, total cholesterol, LDL cholesterol, HDL cholesterol, triglyceride levels)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Atypical Antispychotics (or second generation antipsychotics): Patients with schizophrenia who are currently receiving or are going to start a new treatment with atypical antipsychotics, ziprasidone, risperidone, quetiapine, olanzapine, aripiprazole, amisulpride.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Non-interventional study

SUMMARY:
The purpose of the study is to find and follow-up the metabolic syndrome parameters on patients administering atypical antipsychotics.

DETAILED DESCRIPTION:
Sampling Method Details: Group of patients using the same atypical anti-psychotic.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients diagnosed as schizophrenia by the Diagnostic and Statistical Manual of Mental Disorders.
* Age between 18-45 years
* Patients who started atypical antipsychotic drug treatment or patients who switched from the previous conventional or atypical antipsychotic treatment to another atypical antipsychotic drug treatment by the decision of their physicians.

Exclusion Criteria:

* Patients who are pregnant or considering pregnancy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: * Female and male patients diagnosed as schizophrenia by DSM-IV criteria; Age between 18-45 years
  * Patients who started atypical antipsychotic drug treatment or patients who switched from the previous conventional or atypical antipsychotic treatment to another atypical antipsychotic drug treatment by the decision of their physicians in psychiatry clinics in state and university hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2007-10-23 (Actual); Primary Completion 2008-07-30 (Actual); Study Completion 2008-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- Turkey (Türkiye) (44):
  - Adana Psychiatry and Neurology Hospital, Kurttepe, Adana
  - Pfizer Investigational Site, Kurttepe, Adana
  - Adana Psychiatry and Neurology Hospital, Adana
  - Cukurova University Scool of Medicine, Adana
  - Pfizer Investigational Site, Adana
  - Ankara Oncology Research and Training Hospital, Ankara
  - Pfizer Investigational Site, Ankara
  - Ankara Diskapi Training and Research Hospital, Ankara
  - Ankara Numune Research Hospital, Ankara
  - Ankara Numune Training and Research Hospital Department of Psychiatry, Ankara
  - Antakya Mustafa Kemal University School of Medicine, Antakya
  - Pfizer Investigational Site, Antakya
  - Bolu Psychiatry and Neurology Hospital, Bolu
  - Pfizer Investigational Site, Bolu
  - Pamukkale University School Of Medicine, Denizli
  - Pfizer Investigational Site, Denizli
  - Elazig Mental Illness And Diseases Hospital, Elâzığ
  - Pfizer Investigational Site, Elâzığ
  - Eskisehir Osmangazi University, Eskişehir
  - Pfizer Investigational Site, Eskişehir
  - Bakirkoy Psychiatry and Neurology Hospital, Istanbul
  - Pfizer Investigational Site, Istanbul
  - Bakirkoy Mental Health Hospital, First Clinic of Neurosis, Istanbul
  - Cerrahpasa School of Medicine, Istanbul
  - Erenkoy Psychology and neurology hospital, Istanbul
  - Istanbul University Istanbul School of Medicine, Istanbul
  - Marmara School of Medicine, Istanbul
  - Sisli Etfal Research and training Hospital, Istanbul
  - Vakif Gureba Hospital, Department of Psychiatry, Istanbul
  - Ege University School Of Medicine, Izmir
  - Pfizer Investigational Site, Izmir
  - Kayseri Public Hospital, Kayseri
  - Pfizer Investigational Site, Kayseri
  - Pfizer Investigational Site, Konya
  - Selcuk University Medical School Department of Psychiatry, Konya
  - Manisa Mental Illness And Diseases Hospital, Manisa
  - Pfizer Investigational Site, Manisa
  - 19 may University School of Medicine, Samsun
  - Pfizer Investigational Site, Samsun
  - Samsun Mental Illness And Diseases Hospital, Samsun
  - Pfizer Investigational Site, Trabzon
  - Trabzon Numune Research Hospital, Trabzon
  - Pfizer Investigational Site, Trakya
  - Trakya University School of Medicine, Trakya

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281160&StudyName=An%20Observational%20Study%20On%20Metabolic%20Syndrome%20Parameters%20In%20Schizophrenia%20Patients%20Treated%20With%20Atypical%20Antipsychotics

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects diagnosed with schizophrenia who have been using or recommended to use atypical antipsychotic drugs.
Groups:
- Atypical Antipsychotic Treatment: Subjects with schizophrenia treated with the atypical antipsychotic drugs ziprasidone, risperidone, quetiapine, olanzapine, aripiprazole, or amisulpride. The requirements of the study did not include inducement for any specific atypical antipsychotic drug. The most appropriate treatment for each subject was decided freely by their doctors.
Period: Overall Study
Arm/Group | Atypical Antipsychotic Treatment
Started | 328
Completed | 301 (Number of patients who remained on same medication to end of study.)
Not Completed | 27

BASELINE CHARACTERISTICS:
Arm/Group | Atypical Antipsychotic Treatment
Number analyzed (Participants) | 328
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206
  Male | 122
Region of Enrollment [Number; unit: participants]
  Turkey | 328

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Syndrome Parameter Body Mass Index (BMI)
Description: Iterative mean Body Mass Index at time points.
Time Frame: Baseline, 1 Month, 4 Months
Population: Population : Full Analysis Set. Number of participants analyzed includes subjects with data for each visit.
Measure: Mean (Standard Deviation); unit: kg/m*m (kilograms per meter squared)
Arm/Group | Atypical Antipsychotic Treatment
Number analyzed (Participants) | 163
kg/m*m (kilograms per meter squared)
  Baseline | 26.3 (16.7)
  1 Month | 26.6 (16.3)
  4 Months | 26.9 (17.8)
Statistical Analysis 1: Comparison: Atypical Antipsychotic Treatment; We hypothesize that atypical antipsychotic therapy effects the metabolic syndrome parameters, particularly body mass index; Test type: Superiority or Other; p < 0.001, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant

2. Secondary Outcome: Metabolic Syndrome Parameter BMI by Treatment Group
Description: Iterative measurement of BMI. Mean at time points.
Time Frame: Baseline, 1 Month, 4 Months
Population: Population : Full Analysis Set. Number of participants analyzed includes subjects with data for each visit.
Measure: Mean (Standard Deviation); unit: kg/m*m
Groups:
- Ziprasidone: ziprasidone as prescribed by subject's physician
- Risperidone: risperidone as prescribed by subject's physician
- Quetiapine: quetiapine as prescribed by subject's physician
- Olanzipine: olanzipine as prescribed by subject's physician
- Aripiprazole: aripiprazole as prescribed by subject's physician
- Amisulpride: amisulpride as prescribed by subject's physician
- Other: other medications not included in the protocol-specified atypical antipsychotic groups: clozapine, haloperidol, zuclopenthixol, sertindole, and sulpiride. Treatment prescribed by subject's physician.
Arm/Group | Ziprasidone | Risperidone | Quetiapine | Olanzipine | Aripiprazole | Amisulpride | Other
Number analyzed (Participants) | 25 | 31 | 12 | 33 | 27 | 19 | 16
kg/m*m
  Baseline | 26.12 (18.21) | 26.17 (17.93) | 26.94 (19.82) | 24.06 (18.04) | 29.76 (16.78) | 24.92 (18.25) | 26.41 (16.72)
  1 Month | 26.10 (17.28) | 26.52 (18.65) | 27.70 (20.15) | 24.81 (19.05) | 29.39 (16.33) | 25.12 (19.43) | 26.93 (16.37)
  4 Months | 26.19 (17.90) | 27.23 (20.08) | 28.41 (21.77) | 25.39 (20.34) | 28.75 (18.34) | 25.88 (20.31) | 27.76 (17.79)
Statistical Analysis 1: Comparison: Ziprasidone; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.490, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 2: Comparison: Risperidone; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p < 0.001, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 3: Comparison: Quetiapine; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.006, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 4: Comparison: Olanzipine; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p < 0.001, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 5: Comparison: Aripiprazole; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.003, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 6: Comparison: Amisulpride; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p < 0.001, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 7: Comparison: Other; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.050, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 8: Comparison: Ziprasidone vs Risperidone; Test type: Superiority or Other; p = 0.0012, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Ziprasidone vs Quetiapine; Test type: Superiority or Other; p = 0.0078, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Ziprasidone vs Olanzipine; Test type: Superiority or Other; p = 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Ziprasidone vs Aripiprazole; Test type: Superiority or Other; p = 0.0133, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Ziprasidone vs Amisulpride; Test type: Superiority or Other; p = 0.0142, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Ziprasidone vs Other; Test type: Superiority or Other; p = 0.0265, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Risperidone vs Quetiapine; Test type: Superiority or Other; p = 0.1613, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: Risperidone vs Olanzipine; Test type: Superiority or Other; p = 0.2644, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: Risperidone vs Aripiprazole; Test type: Superiority or Other; p = 0.000005, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: Risperidone vs Amisulpride; Test type: Superiority or Other; p = 0.7385, Wilcoxon (Mann-Whitney)
Statistical Analysis 18: Comparison: Risperidone vs Other; Test type: Superiority or Other; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 19: Comparison: Quetiapine vs Olanzipine; Test type: Superiority or Other; p = 0.6813, Wilcoxon (Mann-Whitney)
Statistical Analysis 20: Comparison: Quetiapine vs Aripiprazole; Test type: Superiority or Other; p = 0.0024, Wilcoxon (Mann-Whitney)
Statistical Analysis 21: Comparison: Quetiapine vs Amisulpride; Test type: Superiority or Other; p = 0.2237, Wilcoxon (Mann-Whitney)
Statistical Analysis 22: Comparison: Quetiapine vs Other; Test type: Superiority or Other; p = 0.5774, Wilcoxon (Mann-Whitney)
Statistical Analysis 23: Comparison: Olanzipine vs Aripiprazole; Test type: Superiority or Other; p = 0.000001, Wilcoxon (Mann-Whitney)
Statistical Analysis 24: Comparison: Olanzipine vs Amisulpride; Test type: Superiority or Other; p = 0.2502, Wilcoxon (Mann-Whitney)
Statistical Analysis 25: Comparison: Olanzipine vs Other; Test type: Superiority or Other; p = 0.5224, Wilcoxon (Mann-Whitney)
Statistical Analysis 26: Comparison: Aripiprazole vs Amisulpride; Test type: Superiority or Other; p = 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 27: Comparison: Aripiprazole vs Other; Test type: Superiority or Other; p = 0.0002, Wilcoxon (Mann-Whitney)
Statistical Analysis 28: Comparison: Amisulpride vs Other; Test type: Superiority or Other; p = 0.8166, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Metabolic Syndrome Parameter Body Weight
Description: Iterative measurement of body weight. Mean at time points.
Time Frame: Baseline, 1 Month, 4 Months
Population: Population : Full Analysis Set. Number of participants analyzed includes subjects with data for each visit.
Measure: Mean (Standard Deviation); unit: kg (kilogram)
Arm/Group | Atypical Antipsychotic Treatment
Number analyzed (Participants) | 173
kg (kilogram)
  Baseline | 74.27 (43)
  1 Month | 75.06 (46)
  4 Months | 76.18 (46)
Statistical Analysis 1: Comparison: Atypical Antipsychotic Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant

4. Primary Outcome: Metabolic Syndrome Parameter Waist Circumference
Description: Iterative measurement of waist circumference. Mean at timepoints.
Time Frame: Baseline, 1 Month, 4 Months
Population: Population : Full Analysis Set. Number of participants analyzed includes subjects with data for each visit.
Measure: Mean (Standard Deviation); unit: cm (centimeter)
Arm/Group | Atypical Antipsychotic Treatment
Number analyzed (Participants) | 173
cm (centimeter)
  Baseline | 91.92 (14.91)
  1 Month | 92.07 (13.54)
  4 Months | 92.80 (12.99)
Statistical Analysis 1: Comparison: Atypical Antipsychotic Treatment; Friedman's test was used to assess trends over time (Baseline, 1 month, 4 months); Test type: Superiority or Other; p < 0.001, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant

5. Primary Outcome: Metabolic Syndrome Parameter Fasting Blood Sugar
Description: Iterative measurement of fasting blood sugar. Mean at time points.
Time Frame: Baseline, 1 Month, 4 Months
Population: Population : Full Analysis Set. Number of participants analyzed includes subjects with data for each visit.
Measure: Mean (Standard Deviation); unit: mg/dl (miligrams per deciliter)
Arm/Group | Atypical Antipsychotic Treatment
Number analyzed (Participants) | 168
mg/dl (miligrams per deciliter)
  Baseline | 80.82 (24.17)
  1 Month | 77.64 (17.74)
  4 Months | 76.79 (19.85)
Statistical Analysis 1: Comparison: Atypical Antipsychotic Treatment; Friedman's test was used to assess trends over time (Baseline, 1 month, 4 months); Test type: Superiority or Other; p = 0.544, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant

6. Primary Outcome: Metabolic Syndrome Parameter Total Cholesterol
Description: Iterative measurement of total cholesterol. Mean at time points.
Time Frame: Baseline, 1 Month, 4 Months
Population: Population : Full Analysis Set. Number of participants analyzed includes subjects with data for each visit.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Atypical Antipsychotic Treatment
Number analyzed (Participants) | 166
mg/dl
  Baseline | 178.48 (47.83)
  1 Month | 181.81 (52.81)
  4 Months | 179.67 (45.27)
Statistical Analysis 1: Comparison: Atypical Antipsychotic Treatment; Friedman's test was used to assess trends over time (Baseline, 1 month, 4 months); Test type: Superiority or Other; p = 0.245, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant

7. Primary Outcome: Metabolic Syndrome Parameter Low Density Lipoprotein (LDL)
Description: Iterative measurement of LDL. Mean at time points
Time Frame: Baseline, 1 Month, 4 Months
Population: Population : Full Analysis Set. Number of participants analyzed includes subjects with data for each visit.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Atypical Antipsychotic Treatment
Number analyzed (Participants) | 143
mg/dl
  Baseline | 118.71 (38.96)
  1 Month | 122.56 (43.23)
  4 Months | 122.86 (39.21)
Statistical Analysis 1: Comparison: Atypical Antipsychotic Treatment; Friedman's test was used to assess trends over time (Baseline, 1 month, 4 months); Test type: Superiority or Other; p = 0.362, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant

8. Primary Outcome: Metabolic Syndrome Parameter High Density Lipoprotein (HDL)
Description: Iterative measurement of HDL. Mean at time points
Time Frame: Baseline, 1 Month, 4 Months
Population: Population : Full Analysis Set. Number of participants analyzed includes subjects with data for each visit.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Atypical Antipsychotic Treatment
Number analyzed (Participants) | 165
mg/dl
  Baseline | 35.11 (13.24)
  1 Month | 36.99 (16.08)
  4 Months | 35.51 (12.00)
Statistical Analysis 1: Comparison: Atypical Antipsychotic Treatment; Friedman's test was used to assess trends over time (Baseline, 1 month, 4 months); Test type: Superiority or Other; p = 0.176, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant

9. Primary Outcome: Metabolic Syndrome Parameter Triglycerides
Description: Iterative measurement of triglycerides. Mean at time points
Time Frame: Baseline, 1 Month, 4 Months
Population: Population : Full Analysis Set. Number of participants analyzed includes subjects with data for each visit.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Atypical Antipsychotic Treatment
Number analyzed (Participants) | 166
mg/dl
  Baseline | 115.11 (78.88)
  1 Month | 116.46 (72.45)
  4 Months | 127.63 (83.45)
Statistical Analysis 1: Comparison: Atypical Antipsychotic Treatment; Friedman's test was used to assess trends over time (Baseline, 1 month, 4 months); Test type: Superiority or Other; p < 0.001, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant

10. Secondary Outcome: Metabolic Syndrome Parameter Weight by Treatment Group
Description: Iterative measurement of weight. Mean at time points.
Time Frame: Baseline, 1 Month, 4 Months
Population: Population : Full Analysis Set. Number of participants analyzed includes subjects with data for each visit.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Ziprasidone | Risperidone | Quetiapine | Olanzipine | Aripiprazole | Amisulpride | Other
Number analyzed (Participants) | 31 | 31 | 12 | 33 | 28 | 20 | 18
kg
  Baseline | 73.11 (14.10) | 72.39 (12.50) | 76.22 (18.01) | 69.82 (10.72) | 84.26 (20.37) | 70.68 (13.49) | 74.77 (15.17)
  1 Month | 73.04 (14.11) | 73.46 (13.14) | 78.41 (18.09) | 71.97 (10.23) | 83.23 (19.81) | 71.02 (12.96) | 76.47 (15.01)
  4 Months | 73.43 (14.44) | 75.47 (13.37) | 80.43 (17.52) | 73.68 (9.87) | 81.55 (17.24) | 73.45 (13.64) | 78.54 (14.96)
Statistical Analysis 1: Comparison: Ziprasidone; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.524, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 2: Comparison: Risperidone; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p < 0.001, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 3: Comparison: Quetiapine; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.005, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 4: Comparison: Olanzipine; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p < 0.001, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 5: Comparison: Aripiprazole; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.009, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 6: Comparison: Amisulpride; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p < 0.001, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 7: Comparison: Other; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.047, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 8: Comparison: Ziprasidone vs Risperidone; Test type: Superiority or Other; p = 0.0007, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Ziprasidone vs Quetiapine; Test type: Superiority or Other; p = 0.0057, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Ziprasidone vs Olanzipine; Test type: Superiority or Other; p = 0.00009, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Ziprasidone vs Aripiprazole; Test type: Superiority or Other; p = 0.0201, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Ziprasidone vs Amisulpride; Test type: Superiority or Other; p = 0.0095, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Ziprasidone vs Other; Test type: Superiority or Other; p = 0.0386, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Risperidone vs Quetiapine; Test type: Superiority or Other; p = 0.1976, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: Risperidone vs Olanzipine; Test type: Superiority or Other; p = 0.2383, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: Risperidone vs Aripiprazole; Test type: Superiority or Other; p = 0.00002, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: Risperidone vs Amisulpride; Test type: Superiority or Other; p = 0.8297, Wilcoxon (Mann-Whitney)
Statistical Analysis 18: Comparison: Risperidone vs Other; Test type: Superiority or Other; p = 0.9081, Wilcoxon (Mann-Whitney)
Statistical Analysis 19: Comparison: Quetiapine vs Olanzipine; Test type: Superiority or Other; p = 0.7386, Wilcoxon (Mann-Whitney)
Statistical Analysis 20: Comparison: Quetiapine vs Aripiprazole; Test type: Superiority or Other; p = 0.0024, Wilcoxon (Mann-Whitney)
Statistical Analysis 21: Comparison: Quetiapine vs Amisulpride; Test type: Superiority or Other; p = 0.2587, Wilcoxon (Mann-Whitney)
Statistical Analysis 22: Comparison: Quetiapine vs Other; Test type: Superiority or Other; p = 0.6263, Wilcoxon (Mann-Whitney)
Statistical Analysis 23: Comparison: Olanzipine vs Aripiprazole; Test type: Superiority or Other; p = 0.000001, Wilcoxon (Mann-Whitney)
Statistical Analysis 24: Comparison: Olanzipine vs Amisulpride; Test type: Superiority or Other; p = 0.2589, Wilcoxon (Mann-Whitney)
Statistical Analysis 25: Comparison: Olanzipine vs Other; Test type: Superiority or Other; p = 0.5153, Wilcoxon (Mann-Whitney)
Statistical Analysis 26: Comparison: Aripiprazole vs Amisulpride; Test type: Superiority or Other; p = 0.0003, Wilcoxon (Mann-Whitney)
Statistical Analysis 27: Comparison: Aripiprazole vs Other; Test type: Superiority or Other; p = 0.0005, Wilcoxon (Mann-Whitney)
Statistical Analysis 28: Comparison: Amisulpride vs Other; Test type: Superiority or Other; p = 0.8952, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Metabolic Syndrome Parameter Waist Circumference by Treatment Group
Description: Iterative measurement of waist circumference. Mean at time points.
Time Frame: Baseline, 1 Month, 4 Months
Population: Population : Full Analysis Set. Number of participants analyzed includes subjects with data for each visit.
Measure: Mean (Standard Deviation); unit: cm (centimeter)
Arm/Group | Ziprasidone | Risperidone | Quetiapine | Olanzipine | Aripiprazole | Amisulpride | Other
Number analyzed (Participants) | 31 | 31 | 12 | 33 | 28 | 20 | 18
cm (centimeter)
  Baseline | 91.18 (14.62) | 91.55 (13.58) | 93.75 (13.37) | 89.04 (18.95) | 96.64 (15.41) | 88.80 (12.38) | 94.06 (11.53)
  1 Month | 90.42 (15.30) | 93.36 (14.50) | 97.28 (14.60) | 87.57 (9.47) | 96.27 (15.72) | 88.53 (10.83) | 94.89 (11.08)
  4 Months | 90.70 (14.84) | 93.52 (13.64) | 97.18 (14.46) | 89.69 (8.82) | 94.92 (15.17) | 90.34 (11.82) | 97.44 (10.35)
Statistical Analysis 1: Comparison: Ziprasidone; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.197, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 2: Comparison: Risperidone; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.010, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 3: Comparison: Quetiapine; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.012, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 4: Comparison: Olanzipine; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p < 0.001, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 5: Comparison: Aripiprazole; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.282, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 6: Comparison: Amisulpride; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.040, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 7: Comparison: Other; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.004, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 8: Comparison: Ziprasidone vs Risperidone; Test type: Superiority or Other; p = 0.0193, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Ziprasidone vs Quetiapine; Test type: Superiority or Other; p = 0.0065, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Ziprasidone vs Olanzipine; Test type: Superiority or Other; p = 0.0002, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Ziprasidone vs Aripiprazole; Test type: Superiority or Other; p = 0.3172, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Ziprasidone vs Amisulpride; Test type: Superiority or Other; p = 0.0116, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Ziprasidone vs Other; Test type: Superiority or Other; p = 0.0016, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Risperidone vs Quetiapine; Test type: Superiority or Other; p = 0.2600, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: Risperidone vs Olanzipine; Test type: Superiority or Other; p = 0.2309, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: Risperidone vs Aripiprazole; Test type: Superiority or Other; p = 0.0063, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: Risperidone vs Amisulpride; Test type: Superiority or Other; p = 0.8158, Wilcoxon (Mann-Whitney)
Statistical Analysis 18: Comparison: Risperidone vs Other; Test type: Superiority or Other; p = 0.3968, Wilcoxon (Mann-Whitney)
Statistical Analysis 19: Comparison: Quetiapine vs Olanzipine; Test type: Superiority or Other; p = 0.7193, Wilcoxon (Mann-Whitney)
Statistical Analysis 20: Comparison: Quetiapine vs Aripiprazole; Test type: Superiority or Other; p = 0.0127, Wilcoxon (Mann-Whitney)
Statistical Analysis 21: Comparison: Quetiapine vs Amisulpride; Test type: Superiority or Other; p = 0.2351, Wilcoxon (Mann-Whitney)
Statistical Analysis 22: Comparison: Quetiapine vs Other; Test type: Superiority or Other; p = 0.5672, Wilcoxon (Mann-Whitney)
Statistical Analysis 23: Comparison: Olanzipine vs Aripiprazole; Test type: Superiority or Other; p = 0.00009, Wilcoxon (Mann-Whitney)
Statistical Analysis 24: Comparison: Olanzipine vs Amisulpride; Test type: Superiority or Other; p = 0.1774, Wilcoxon (Mann-Whitney)
Statistical Analysis 25: Comparison: Olanzipine vs Other; Test type: Superiority or Other; p = 0.6082, Wilcoxon (Mann-Whitney)
Statistical Analysis 26: Comparison: Aripiprazole vs Amisulpride; Test type: Superiority or Other; p = 0.0079, Wilcoxon (Mann-Whitney)
Statistical Analysis 27: Comparison: Aripiprazole vs Other; Test type: Superiority or Other; p = 0.0014, Wilcoxon (Mann-Whitney)
Statistical Analysis 28: Comparison: Amisulpride vs Other; Test type: Superiority or Other; p = 0.5587, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Metabolic Syndrome Parameter Triglycerides by Treatment Group
Description: Iterative measurement of triglycerides. Mean at time points.
Time Frame: Baseline, 1 Month, 4 Months
Population: Population : Full Analysis Set. Number of participants analyzed includes subjects with data for each visit.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Ziprasidone | Risperidone | Quetiapine | Olanzipine | Aripiprazole | Amisulpride | Other
Number analyzed (Participants) | 28 | 29 | 12 | 33 | 28 | 20 | 16
mg/dl
  Baseline | 104.89 (85.13) | 129.66 (90.13) | 117.92 (80.54) | 86.24 (40.00) | 113.79 (88.12) | 142.75 (83.42) | 131.88 (74.23)
  1 Month | 92.25 (55.81) | 121.00 (78.34) | 141.50 (78.34) | 97.48 (49.76) | 111.78 (82.98) | 133.90 (67.17) | 157.38 (90.16)
  4 Months | 94.04 (45.98) | 148.14 (88.69) | 119.33 (55.21) | 110.97 (52.32) | 127.07 (80.83) | 161.85 (143.26) | 148.00 (81.76)
Statistical Analysis 1: Comparison: Ziprasidone; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.077, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 2: Comparison: Risperidone; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.039, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 3: Comparison: Quetiapine; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.978, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 4: Comparison: Olanzipine; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p < 0.001, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 5: Comparison: Aripiprazole; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.593, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 6: Comparison: Amisulpride; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.987, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant
Statistical Analysis 7: Comparison: Other; Friedman's test was used to assess trends over time; Test type: Superiority or Other; p = 0.174, Friedman — P-value was not adjusted for multiple comparisons; p-values < 0.05 were considered statistically significant

ADVERSE EVENTS:
Arm/Group | Ziprasidone | Risperidone | Quetiapine | Olanzipine | Aripiprazole | Amisulpride | Other
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/64 | 0/23 | 0/60 | 0/50 | 0/41 | 0/33
Other Adverse Events (participants affected / at risk) | 4/57 | 14/64 | 5/23 | 27/60 | 12/50 | 9/41 | 33/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=57) | Risperidone (N=64) | Quetiapine (N=23) | Olanzipine (N=60) | Aripiprazole (N=50) | Amisulpride (N=41) | Other (N=33)
Menstrual irregularities (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Akathisia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 5
Akathisia + sedation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Allergy + Sedation (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Giddiness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspahlgia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dystasia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dystonia (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Epileptic exacerbation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Extrapyramidal syndrome (General disorders) | 0 | 5 | 3 | 3 | 0 | 0 | 27
Hyperprolactinemia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hypertension (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight gain (General disorders) | 2 | 2 | 1 | 12 | 6 | 1 | 0
Weight gain + QT extension (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight gain + Sedation (General disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Leucopenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sedation (General disorders) | 0 | 1 | 1 | 6 | 2 | 1 | 1
Late Dischinesia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2
Tremor (General disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 2
Tremor + Insomnia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.